CLINICAL TRIAL: NCT05894135
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of BG2109 in Chinese Subjects With Endometriosis
Brief Title: Efficacy and Safety of BG2109 in Chinese Subjects With Endometriosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bio Genuine (Shanghai) Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BG2109-AB-301
Record Dates: First submitted 2023-05-09; First posted 2023-06-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Endometriosis; Moderate to Severe Endometriosis-associated Pain
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BG2109 100 mg group (Experimental)
  Interventions: Drug: BG2109 100mg; Drug: BG2109 200mg Placebo; Drug: ABT Placebo
- BG2109 200 mg +ABT group (Experimental)
  Interventions: Drug: BG2109 200mg; Drug: ABT(E2 1 mg / NETA 0.5 mg); Drug: BG2109 100mg Placebo
- Placebo group (Placebo Comparator)
  Interventions: Drug: BG2109 100mg Placebo; Drug: BG2109 200mg Placebo; Drug: ABT Placebo

INTERVENTIONS:
Drug: BG2109 100mg — One tablet of BG2109 100mg , oral , once daily
  Arms: BG2109 100 mg group
Drug: BG2109 200mg — One tablet of BG2109 200mg, oral , once daily.
  Arms: BG2109 200 mg +ABT group
Drug: ABT(E2 1 mg / NETA 0.5 mg) — One tablet of ABT(E2 1 mg / NETA 0.5 mg), oral, once-daily
  Arms: BG2109 200 mg +ABT group
Drug: BG2109 100mg Placebo — One tablet of BG2109 100mg Placebo, oral , once daily.
  Arms: BG2109 200 mg +ABT group; Placebo group
Drug: BG2109 200mg Placebo — One tablet of BG2109 200mg Placebo, oral , once daily.
  Arms: BG2109 100 mg group; Placebo group
Drug: ABT Placebo — One tablet of ABT Placebo, oral, once-daily
  Arms: BG2109 100 mg group; Placebo group

SUMMARY:
The objective of this study is to demonstrate the efficacy and safety of BG2109 administered orally once daily at a dose of 100 mg alone or of 200 mg in combination with add-back hormone replacement therapy (ABT: estradiol (E2) 1 mg / norethisterone acetate (NETA) 0.5 mg) versus placebo, while under randomized treatment, in the management of moderate to severe endometriosis-associated pain (EAP) in chinese women with surgically confirmed endometriosis

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study to demonstrate the efficacy and safety of BG2109 administered orally once daily at doses of 100 mg alone and 200 mg in combination with low dose ABT (E2 1 mg/NETA 0.5 mg) versus placebo in the management of moderate to severe EAP in chinese women with surgically confirmed endometriosis.

The entire study is divided into the core stage and the extension stage, with a total duration of approximately 72 weeks. This includes the prescreening wash-out period (if applicable), screening period (approximately 5-8 weeks), core stage (24 weeks) and extension stage (28 weeks), and the safety follow-up period (approximately 12 weeks)

ELIGIBILITY:
Key Inclusion Criteria:

1. The subject must be a premenopausal woman aged ≥18 years.
2. The subject must have had her most recent surgical and histological diagnosis of pelvic endometriosis (laparoscopy, laparotomy, vaginal fornix or other biopsy) within 10 years and at least 2 months ago prior to screening.
3. The subject has moderate to severe EAP during the screening period defined as:

   1. At the screening visit, a score of at least 2 for DYS and at least 2 for NMPP for the previous month assessed with the modified Biberoglu & Behrman (mB&B) scale
   2. Subject is confirmed to meet the following criteria during the screening period, within 35 consecutive calendar days prior to the baseline visit:

   i. Mean overall pelvic pain scores on the 0-10 NRS over the 5 days with the highest score ≥ 4; ii. At least two days with "moderate" or "severe" pain on the 0-3 VRS for pelvic pain over the days with uterine bleeding; iii. At least two days with "moderate" or "severe" pain on the 0-3 VRS for pelvic pain over the days without uterine bleeding;
4. The subject has a Body Mass Index (BMI) ≥ 18 kg/m2 at the screening visit

Key Exclusion Criteria:

1. The subject is pregnant or breastfeeding, or plans to become pregnant during the study treatment period.
2. The subject has a surgical history of:

   1. Hysterectomy,
   2. Bilateral oophorectomy,
   3. Surgeries that interfere with gastrointestinal motility, pH value, or absorption (including vagotomy, enterectomy, or gastric surgery),
   4. Any major abdominal surgery (including laparotomy for endometriosis) within 6 months or any interventional surgery for endometriosis (i.e. laparoscopy) performed within a period of 2 months before screening, or the subject is scheduled for a surgical abdominal procedure during the course of the study.
3. The subject may need to take prohibited medications during the study or in the stipulated time before screening
4. The subject has a contra-indication to ABT
5. The subject has chronic pelvic pain that, in the opinion of the Investigator, is not caused by endometriosis and requires chronic analgesic or other chronic therapy which would interfere with the assessment of EAP
6. The subject has conditions that affect bone mass density (BMD) assessment
7. The subject did not respond to prior treatment with GnRH agonists or GnRH antagonists for endometriosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dysmenorrhea (DYS) response rate at Week 12 | Week 12
  responders are defined as those with a significant decrease in mean DYS score measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse) compared to baseline, with decreased or stable analgesic use for EAP
Non-menstrual pelvic pain (NMPP) response rate at Week 12 | Week 12
  responders are defined as those with a significant decrease in mean NMPP score measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse) compared to baseline, with decreased or stable analgesic use for EAP

SECONDARY OUTCOMES:
Change of the interference of pain with the ability to perform daily activities from the baseline at week 24 | Week 24
  measured using the pain dimension in Endometriosis Health Profile-30 (EHP-30)(0-100, higher scores mean worse)
Change of the mean overall pelvic pain(OPP) score from the baseline at week 24 | Week 24
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of the mean DYS score from the baseline at week 24 | Week 24
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of the mean NMPP score from the baseline at week 24 | Week 24
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Ratio of subjects who do not use analgesics to treat EAP at week 24 | Week 24

OTHER OUTCOMES:
Change of mean pelvic pain scores of DYS from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of mean pelvic pain scores of NMPP from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of mean pelvic pain scores of overall pelvic pain(OPP) from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of mean scores of dyschezia from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of mean scores of dyspareunia from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using Verbal rating scale - VRS(0-3, higher scores mean worse)
Change of the number of days with moderate to severe pelvic pain from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of the number of days with uterine bleeding (including spotting) from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using the uterine bleeding scale(0-3, higher scores mean worse)
Change of the number of days of analgesic use (including any class) for EAP from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
Change of the mean worst pelvic pain score defined as the mean of the 5 highest daily pain scores from the baseline to each scheduled assessment | during the previous 35 days of Week 4,8,12,24,28,32,36,52,56,64
  measured using Numeric Rating Scale - NRS(0-10, higher scores mean worse)
Change of scores in the dimensions of pain, control and powerlessness, emotional well-being, social support, self-image, and sexual relationships from the baseline to each scheduled assessment | during the previous 28 days of Week 4,8,12,24,36,52,56,64
  measured using the EHP-30 core questionnaire（contains 5 dimensions：pain, control and powerlessness, emotional well-being, social support, self-image; all are 0-100 score, higher scores mean worse） and Module C（0-100 score, higher scores mean worse）
Change of score of quality of life from the baseline to week 24 and week 52 | during the previous 28 days of Week 24,52,
  measured using SF-36v2 ® Health Survey (SF-36v2)（0-100 score, higher scores mean better ）
Change of uterine size of a patient with concomitant adenomyosis from the baseline to week 12, week 24, and week 52 | Week 12,24,52
Change of BMD on lumbar (L1-L4), femoral neck, and total hip from the baseline to week 24 and week 52 | Week 24,52
  measured using dual-energy x-ray absorptiometry (DXA)
Incidence and severity of treatment emergent adverse events (TEAEs) during treatment period | from first dose to Week 52
Incidence and severity of hypoestrogenic TEAEs (vasomotor symptoms) | from first dose to Week 52
Time to the first post-treatment menses | Week 56 or 64

CONTACTS AND LOCATIONS:
Overall Officials: Congjian Xu, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics & Gynecology Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No